CLINICAL TRIAL: NCT00932633
Title: Role of Inflammatory Response in Brain Injury Following Neonatal Cardiac Surgery
Brief Title: Magnetic Resonance Imaging (MRI) to Evaluate Brain Injury in Congenital Heart Disease
Acronym: CHD Brain
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, William T. Mahle, MD, Associate Professor, Emory University
Other Study IDs: IRB00017965; 17965 (Other: Other)
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Neonatal Congenital Heart Disease
Keywords: neonatal brain injury; congenital heart disease; magnetic resonance imaging; cardiopulmonary bypass; neurodevelopmental outcome
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — dried blood spot sample
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Infants with congenital heart disease (CHD) requiring surgery frequently have brain injury seen on magnetic resonance imaging (MRI). This occurs in approximately 40% of these newborns, and even though these are full-term infants, the injury seen closely resembles the same form of brain injury that can be seen in premature babies. Much like premature newborns, infants with CHD also have long-term neurodevelopmental problems (in over 50%).

The investigators do not know why infants with CHD get this specific form of brain injury. One risk factor is felt to be the inflammation that occurs in response to heart-lung bypass (cardiopulmonary bypass, or CPB), a necessary feature of open-heart surgery. Newborns have a stronger inflammatory reaction to CPB than older children or adults. The investigators do know from animal experiments and other human data that inflammation can be harmful to the developing brain.

The investigators hypothesize that children with CHD requiring surgery as a newborn have brain injury due to toxicity from the inflammatory response. The investigators will test this by enrolling newborns undergoing heart surgery to measure markers of inflammation, measure brain injury by MRI, and then test their developmental outcome at 1 and 2 years of age.

An association between inflammation and injury might impact what medicines are chosen to protect the brain in future studies, even in other populations such as preterm infants.

DETAILED DESCRIPTION:
Term infants with congenital heart disease (CHD) requiring neonatal surgery have an unusual susceptibility to white matter injury (WMI), a neuropathology typically seen in preterm infants. The mechanism of this brain injury is unclear. Newborns with CHD may experience a dramatic peri-operative inflammatory response during critical periods of neurodevelopment. Experimental models suggest certain pro-inflammatory cytokines can be toxic to developing oligodendrocytes, resulting in white matter pathology. The consequence of exposure to the systemic inflammatory response (SIR) in this group of patients is unknown; however, neuroimaging abnormalities (seen in approximately 40%) and neurodevelopmental impairment (noted in approximately 50%) are both well established in children with CHD. We hypothesize that term newborns with complex CHD requiring neonatal surgery have WMI due to neurotoxicity from the profound peri-operative inflammatory response. These hypotheses will be tested in a prospective longitudinal study that will characterize the SIR (Aim 1) in a heterogeneous group of congenital lesions/surgeries, assess brain injury in the post-operative period (Aim 2), asses neurodevelopment outcomes at 1 and 2 years (Aim 3), and determine whether inflammation plays a mechanistic role (Aim 2a, 3a).

ELIGIBILITY:
Inclusion Criteria:

* Term or near-term (> 35 week gestation) neonates with CHD presenting for cardiac surgery
* Less than 30 days old
* No patient will be excluded because of race or ethnicity
* Parental or legal guardian consent will be obtained for all patients prior to enrollment

Exclusion Criteria:

* Newborns with multiple organ abnormalities in addition to their heart defect such as diaphragmatic hernia, tracheo-esophageal fistula, and congenital syndromes will be excluded from participation
* Newborns with either genetic syndromes or congenital infections that are associated with developmental delay will also be excluded
* Newborns with perinatal depression as defined by a cord blood gas pH < 7.0 or a 5 minute Apgar score < 5, will be excluded
* Patients with multiple organ failure, syndromes, and perinatal depression have other causes for neurodevelopmental abnormalities
* Those patients unable to return for postoperative follow-up and neurodevelopmental testing will also be excluded from participation
* Parent or legal guardian unable or unwilling to consent
* Non-English speaking families

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: newborns with congenital heart disease requiring surgery during the first 30 days of life
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2009-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be a measure of the association of pro-inflammatory cytokines with WMI score | 5 years

SECONDARY OUTCOMES:
Association between inflammatory response and neurodevelopmental testing | 5 years
Association of neuroimaging abnormalities with neurodevelopmental testing | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: William T Mahle, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided